CLINICAL TRIAL: NCT05077969
Title: A Virtual Phase 2 Randomized, Placebo-controlled, Double-blind Study to Evaluate the Safety and Efficacy of the Combination of Famotidine and Celecoxib as a Post-exposure Prophylaxis (PEP) for Newly-infected COVID-19 Patients
Brief Title: Leidos-Enabled Adaptive Protocol (LEAP-CT) for Evaluation of Post-exposure Prophylaxis for Newly-infected COVID-19 Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Leidos Life Sciences (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LDOS-21-001-02
Record Dates: First submitted 2021-10-07; First posted 2021-10-14 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: 2019 Novel Coronavirus Disease; 2019 Novel Coronavirus Infection; 2019-nCoV Disease; 2019-nCoV Infection; COVID-19; COVID-19 Pandemic; COVID-19 Virus Disease; COVID-19 Virus Infection; Covid19; Coronavirus Disease 2019; SARS-CoV2 Infection; SARS-CoV-2 Acute Respiratory Disease
Keywords: COVID-19; COVID; COVID19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Famotidine; Celecoxib

STUDY DESIGN:
Intervention Model Description: Participants randomized 1:1, study drug:placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Study Product) (Experimental): Participants will receive 80 mg famotidine (PO) QID and 400 mg celecoxib as a first dose, followed by 200 mg (PO) BID celecoxib, for 5 days. Following this 5-day period, participants will continue their famotidine treatment for an additional 9 days.
  Interventions: Drug: Famotidine; Drug: Celecoxib
- Group 2 (Reference Therapy) (Placebo Comparator): Participants will receive matching placebos QID and BID, for 5 days. Following this 5-day period, participants will continue to receive matching famotidine placebo, QID, for an additional 9 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Famotidine — 80 mg tablet, QID for 14 days
  Other Names: Pepcid
  Arms: Group 1 (Study Product)
Drug: Celecoxib — 400 mg (initial dose), then 200 mg capsule, BID for 5 days
  Other Names: Celebrex
  Arms: Group 1 (Study Product)
Drug: Placebo — tablet, QID for 14 days; capsule, BID for 5 days
  Arms: Group 2 (Reference Therapy)

SUMMARY:
This study is designed to test the efficacy and safety of combinations of two well-understood agents - famotidine and celecoxib. Each of these agents separately demonstrate clinical activity in mitigating COVID-19 disease symptoms or severity, and each of which appear to have separate and complementary mechanisms of action.

DETAILED DESCRIPTION:
Qualifying patients will have been confirmed positive for COVID-19 and have symptoms of World Health Organization (WHO) Ordinal Scale for Clinical Improvement with scores of ≤3 on the 11-point scale and will be randomly assigned, in a 1:1 ratio, to one of two regimens, with 659 participants per group, as follows:

Group 1 (study product) participants will receive 80 mg famotidine by mouth (PO) 4 times per day (QID) + 400 mg celecoxib as a first dose, followed by 200 mg celecoxib (PO) 2 times per day (BID), for 5 days. Following this 5-day period, participants will continue their famotidine treatment for an additional 9 days.

Group 2 (reference therapy) participants will receive matching placebos QID and BID, for 5 days. Following this 5-day period, participants will continue to receive matching famotidine placebo, QID, for an additional 9 days.

Safety and efficacy of famotidine and celecoxib will be evaluated.

This is a completely virtual trial and you can participate from your own home. Please call 1-888-370-9330 to speak to someone regarding study participation in your area.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants must be at least 18 years of age, inclusive, at the time of signing the informed consent form.
* Confirmed SARS-CoV-2 polymerase chain reaction (PCR) positive patient within 5 days of enrollment, as shown by medical history and reported PCR test result.
* Reports having one or more symptoms consistent with SARS-CoV-2, as defined in Master Protocol Appendix 3 Table 4.
* COVID-19 diagnosis must be WHO grade ≤3.
* Contraceptive use by men or women should be consistent with Appendix 4 of the Master protocol (LDOS-21-001).
* Reliable access to the Internet via a browser installed on personal device or computer.
* Capable of understanding and providing signed informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Ongoing antiviral or antiretroviral treatment
* Known history of HIV
* Ongoing anti-inflammatory treatment that cannot be temporarily discontinued during the study. This includes nonsteroidal anti-inflammatory drugs (NSAIDs), and corticosteroids - including Dexamethasone (dexamethasone administration restricted to recommended standard of care use per NIH COVID-19 Guidelines)

  1. drugs dependent on gastric pH for absorption, e.g., dasatinib, delavirdine, mesylate, cefditoren, and fosamprenavir;
  2. tizanidine (CYP1A2) substrate;
  3. drugs that interfere with hemostasis (e.g., warfarin, aspirin, selective serotonin reuptake inhibitors [SSRIs]/serotonin norepinephrine reuptake inhibitors (SNRIs]);
  4. angiotensin converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARB), or beta-blockers;
  5. diuretics;
  6. digoxin
* Ongoing treatment that cannot be temporarily discontinued during the study, with: antimalarials, antiarrhythmics, tricyclic antidepressants, natalizumab, quinolones, macrolides, agalsidase alfa and beta
* Ongoing famotidine or celecoxib or other COVID-19 clinical investigational treatment(s) within the past 30 days, or current participation in another investigational clinical trial
* History of asthma, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDs
* History of immunosuppression
* Rejection of participation by Principal Investigator or Sponsor
* Any contraindication for famotidine or celecoxib treatment:

  1. Famotidine or celecoxib hypersensitivity
  2. Retinopathy, visual field or visual acuity disturbances
  3. History of cardiovascular disease, such as congestive heart failure, QT prolongation, myocardial infarction, bradycardia (<50 bpm), ventricular tachycardia, other arrhythmias
  4. Myasthenia gravis
  5. Psoriasis or porphyria
  6. History of renal failure/dialysis or a glomerular clearance <60 mL/min
  7. History of severe hypoglycemia
  8. Moderate or severe hepatic impairment, e.g., Child-Pugh Class B or C
  9. Known or suspected to be poor CYP2C9 metabolizers based on genotype or previous history or experience with other CYP2C9 substrates, such as warfarin and phenytoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Roberts, MS, PMP, Study Director — Leidos, Inc.
Locations (15):
- United States (15):
  - Integrated Therapeutic Solutions USA, Inc., Newport Beach, California
  - Integrated Therapeutic Solutions USA, Inc., Miami, Florida
  - Integrated Health Solutions USA, Inc., Atlanta, Georgia
  - Integrated Therapeutic Solutions USA, Inc, Hazlehurst, Georgia
  - Integrated Therapeutic Solutions USA, Inc., Chicago, Illinois
  - Integrated Therapeutic Solutions USA, Inc, Prospect, Kentucky
  - Integrated Therapeutic Solutions USA, Inc, Frederick, Maryland
  - Integrated Therapeutic Solutions USA, Inc, Gaithersburg, Maryland
  - Integrated Therapeutic Solutions USA, Inc, Rockville, Maryland
  - Integrated Therapeutic Solutions USA, Inc, Dearborn, Michigan
  - Integrated Therapeutic Solutions USA, Inc., Newark, New Jersey
  - Integrated Therapeutic Solutions USA, Inc., New York, New York
  - Integrated Therapeutic Solutions USA, Inc., Huntingdon, Pennsylvania
  - Integrated Therapeutic Solutions USA, Inc., Charleston, South Carolina
  - Integrated Therapeutic Solutions USA, Inc., Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make individual participant data (IPD) available.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 9 patients were randomized into the study only 4 patients received study drug due to early termination of the study.
Period: Overall Study
Arm/Group | Group 1 (Study Product) | Group 2 (Reference Therapy)
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Study Product) | Group 2 (Reference Therapy) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 42.5 [40 to 45] | 27 [26 to 28] | 34.75 [26 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With at Least One COVID-19-related Medically Attended Contact Due to Increased COVID-19 Symptom Severity
Description: Medically attended contact will be measured in whole numbers and reported as "1 medically attended contact" each time, in the electronic data capture system for all study participants.
Time Frame: Through Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Study Product) | Group 2 (Reference Therapy)
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

2. Primary Outcome: Number of Patients With at Least One COVID-19-related Medically Attended Contact Due to Death (All-cause Mortality).
Description: Medically attended contact will be measured in whole numbers and reported as "1 medically attended contact" in the electronic data capture system for all study participants.
Time Frame: Through Day 30
Population: Participants were all white (non-Hispanic) females between 18 and 65 years of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Study Product) | Group 2 (Reference Therapy)
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (SAE) as Assessed by Participant Withdrawal
Description: Study discontinuation will be measured in whole units, by number of participants who are removed with the reason of "SAE" and captured by the electronic data capture system.
Time Frame: 90 days
Population: Participants were all white (non-Hispanic) females between 18 and 65 years of age.
Measure: Number; unit: participants
Arm/Group | Group 1 (Study Product) | Group 2 (Reference Therapy)
Number analyzed (Participants) | 1 | 2
participants | 0 | 0

4. Secondary Outcome: Incidence of Death
Description: Deaths will be captured by whole numbers, by number of participants who are removed from the study with reason as "death" in the electronic data capture system.
Time Frame: 90 days
Population: Participants were all white (non-Hispanic) females between 18 and 65 years of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Study Product) | Group 2 (Reference Therapy)
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Group 1 (Study Product) | Group 2 (Reference Therapy)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Study Product) (N=2) | Group 2 (Reference Therapy) (N=2)
Sinus Headaches (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was not able to enroll the requisite number of patients to evaluate the prespecified endpoints. As a result the study was halted prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT05077969/Prot_000.pdf
  • Informed Consent Form (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT05077969/ICF_001.pdf